CLINICAL TRIAL: NCT02892617
Title: Evaluation of the Prevalence of Germs Slow Growth in the Intervertebral Disc (IVD) During Spinal Surgery: a Single-center Prospective Observational Study
Brief Title: Evaluation of the Prevalence of Germs Slow Growth in the Intervertebral Disc (IVD) During Spinal Surgery
Acronym: DISCO-PROP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-A01831-44
Record Dates: First submitted 2016-08-25; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-08

CONDITIONS: Prevalence of Germs; Spinal Surgery; Anterior Disc Disease; Modic 1
Keywords: Modic 1; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Disc
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients with low back pain lasting for more than 6 months, debilitating, with the presence of type 1 Modic disc disease on MRI at the operated disc, eligible for a disc prosthesis or arthrodesis anterior approach
  Interventions: Other: Bacteriological analysis of disc
- Group 2: Patients underwent surgery for nerve root pain by disc herniation on MRI viewable with a radio-clinical concordance with or without Modic 1 disc disease in the operated disc
  Interventions: Other: Bacteriological analysis of disc

INTERVENTIONS:
Other: Bacteriological analysis of disc

SUMMARY:
Low back pain is one of the most frequent reasons for consultation in rheumatology. There is a strong correlation between low back pain, and the presence of a type of Modic 1 signal on MRI.

The anomaly Modic 1 results in a hypointense signal T1-weighted images and hyperintense on T2-weighted sequences (including T2 STIR and / or Fat Sat) and contrast enhancement of the endplates after gadolinium injection; it corresponds to a replacement of normal cancellous bone of fibrovascular tissue.

The origin of this inflammatory process Modic 1 into the vertebra is still unknown.

infectious hypothesis was raised, including contamination by germs called "slow-growth" such as Propionibacterium acnes (PA).

Many studies interesting Bacteriological analysis of disc material found the presence of bacteria (prevalence between 0 and 54%).

A recent clinical trial evaluating the efficacy of antibiotic treatment compared to placebo in low back pain with Modic 1; a show effectiveness of this treatment on the different clinical parameters evaluated.

However skin contamination is not formally excluded, particularly in patients previously infiltrated (including epidural).

Our hypothesis is that the slow-growing bacteria are not involved in Modic 1 type of disc disease, and the possible presence of PA or other slow-growing bacteria in samples obtained discal posterior approach would be related to intraoperative contamination or during preoperative spinal infiltrations The main objective is to assess the prevalence of germs slow growth in the intervertebral disc in the spinal surgery by anterior disc disease in type 1 Modic.

ELIGIBILITY:
Inclusion Criteria:

* Major patients accepted to participate in the study and who signed an informed consent.
* Patients with low back pain lasting for more than 6 months, disabling, with disc disease type 1 Modic eligible for a disc prosthesis or arthrodesis anterior approach.
* Patients underwent surgery for nerve root pain by disc herniation on MRI viewable with a radio-clinical concordance with or without Modic 1 disc disease in the operated disc

Exclusion Criteria:

* Lumbar spine surgery history within 12 months and / or presence of osteosynthesis material.
* Immunocompromised patients (HIV, cancer, immunosuppressive treatment, lupus, chronic infection, ...)
* Patients previously treated with antibiotics exceeding 15 days during last 3 months prior enrollment for a period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Disc samples taken during spine surgery during installation of disc prostheses or inter somatic cages made by anterior approach in type discopathies Modic.
  Fragments disc withdrawn during cures herniated disc surgeries by posterior way.
  Patients were recruited from the orthopedic service and Neurosurgery at Henri Mondor Hospital in Creteil
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Presence or lack of germs slow growth in disc by standard culture and molecular biology technique (16S RNA). | Visit 2 (surgery day)

CONTACTS AND LOCATIONS:
Locations (1):
- Henri Mondor Hospital, Créteil, France